CLINICAL TRIAL: NCT01836562
Title: A Clinical Trial to Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Autism. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: A Clinical Trial to Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Autism
Acronym: BMCA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00105
Record Dates: First submitted 2013-02-26; First posted 2013-04-22 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Autism
Keywords: Autism stem cell MNCs
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STEM CELL (Other): intra thecal injection of MNC stem cell therapy
  Interventions: Biological: STEM CELL THERAPY

INTERVENTIONS:
Biological: STEM CELL THERAPY — Intra thecal injection of autologous MNC ,Intra thecal inj.of 100 millions MNC in 3 doses at 10 days interval.
  Other Names: Intra thecal injection of autologous MNC

SUMMARY:
This clinical trial is a single Arm, single centre to check the safety and efficacy of bone marrow derived autologous mono nuclear cells (MNC) (100 million per dose). Trial to be conducted for 36 months.

DETAILED DESCRIPTION:
Autism is a developmental disorder that appears in the first 3 years of life, and affects the brain's normal development of social and communication skills. Autism is a physical condition linked to abnormal biology and chemistry in the brain. The exact causes of these abnormalities remain unknown,Symptoms-Children with autism typically have difficulties in: Pretend play, Social interactions, Verbal and non-verbal communication. Some children with autism appear normal before age 1 or 2 and then suddenly "regress" and lose language or social skills they had previously gained. This is called the regressive type of autism. People with autism may: Be overly sensitive in sight, hearing, touch, smell, or taste.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from Autism.
* willingness to undergo bone marrow derived autologous cell therapy.
* patient those provide fully Informed consent form for the study.
* Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.

Exclusion Criteria:

* Patients with pre - existing or Current systemic disease such as lung , liver ( exception; History of uncomplicated Hepatitis A),gastrointestinal, Cardiac , Immunodeficiency,(including HIV) Or laboratory Investigation that could cause a neurological defect.History of Life threatening Allergic or immune- mediated reaction.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in childhood autism rating scale | 6 month

SECONDARY OUTCOMES:
Improvement in perfusion of brain with PET scan report | 6 MONTH

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India